CLINICAL TRIAL: NCT05721547
Title: Alterations in Spinal Alignment and Mobility in Individuals With Arthroscopic Rotator Cuff Repair: Which Factors Differ From Healthy Individuals?
Brief Title: Alterations in Spinal Alignment and Mobility in Individuals With Arthroscopic Rotator Cuff Repair
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Beyza Yazgan Dagli, Research Assistant, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-BYD-02
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Rotator Cuff Tears; Posture; Spinal Curvatures; Arthroscopic Surgery
MeSH Terms: conditions — Rotator Cuff Injuries; Spinal Curvatures | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RC Repair Group: Participants who had undergone the same arthroscopic RM surgical procedure and technique; had undergone acromioplasty and/or tenodesis with RM repair; had undergone arthroscopic RM surgery from the upper extremity of the dominant side; had completed six months following surgery
  Interventions: Other: Assessment
- Healthy Group: Participants who had not undergone any shoulder surgery, had no history of shoulder-related pain, discomfort, or trauma in the last year
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Assessment

SUMMARY:
The aim of this observational study was to the alterations in spinal alignment in individuals who have undergone RC surgery and revealed the differences compared to healthy individuals.

DETAILED DESCRIPTION:
Shoulder dysfunctions are thought to be predisposed by poor posture and muscle imbalances. The shoulder functionality could be limited or worsened by a restricted range of motion (ROM) of the spine. Evidence from studies evaluating both people with shoulder pain and asymptomatic participants indicates a relationship between a decreased thoracic kyphosis and an increased shoulder ROM. Therefore, a higher thoracic kyphosis may be linked to a lower ROM in the shoulder. Shoulder dysfunction becomes more common after the age of 40, and the relationship between spinal posture and shoulder dysfunction is crucially needed to be assessed.

The aim of this observational study was to the alterations in spinal alignment and mobility in individuals who have undergone RC surgery and revealed the differences compared to healthy individuals.

This cross-sectional observational study was conducted with patients who underwent arthroscopic RM surgery and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* those who had undergone the same arthroscopic RM surgical procedure and technique
* had undergone acromioplasty and/or tenodesis with RM repair
* had undergone arthroscopic RM surgery from the upper extremity of the dominant side;
* had completed six months following surgery; were able to perform active shoulder elevation movements of 90° or more
* were between the ages of 40 and 75
* were volunteers to participate in the study.

Exclusion Criteria:

* who had undergone previous shoulder surgery or revision surgery, subscapularis tendon repair in addition to RM repair, scoliosis surgery, or any surgeries to limit spine motion, as well as those with a history of upper extremity fractures, diabetes mellitus, hypertension, cardiovascular disease, or chronic respiratory diseases that could limit the test's ability to be accomplished

Ages: 40 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent arthroscopic RM surgery who had undergone the same arthroscopic RM surgical procedure and technique
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Spinal alignment and mobility assessment | 8 months
  The Spinal Mouse (IDIAG M360), novel, a computer-aided electronic measuring tool that noninvasively evaluates spinal range of motion and intersegmental angles, was used to examine spinal posture. The Spinal Mouse device is reliable and valid for the assessment of spine mobility and posture

SECONDARY OUTCOMES:
Scapular dyskinesia | 8 months
  Performed using the observational scapular dyskinesia test
Range of Motion | 8 months
  Performed using with Goniometer
Postural stability | 8 months
  Performed using with functional reach test

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided